CLINICAL TRIAL: NCT04750967
Title: Comparison of Amitriptyline and Nerve Blocks (GON and SON) in Patients With Migraine
Brief Title: Amitriptyline vs GON and SON Blocks in Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cem Bölük, Principal Investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-70847213-929-3410
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Migraine; Headache
Keywords: greater occipital nerve; supraorbital nerve; nerve blocks
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Lidocaine; Amitriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Greater occipital nerve and supraorbital nerve block with 1% lidocaine once a week for first four weeks then once a month for 5 months
  Interventions: Drug: Lidocaine 1% Injectable Solution
- Control (Active Comparator): Amitriptyline 25 mg daily for 6 months
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Lidocaine 1% Injectable Solution — Repeated injections of lidocaine to greater occipital nerve and supraorbital nerve once a week for first four weeks then once a month for five months
  Arms: Active
Drug: Amitriptyline — Amitriptyline 25 mg daily
  Arms: Control

SUMMARY:
Comparison of efficacy and safety of amitriptyline and nerve blocks

DETAILED DESCRIPTION:
This study aims to compare the efficacy and safety of amitriptyline and nerve blocks (greater occipital nerve and supraorbital nerve)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with migraine according to ICHD-3

Exclusion Criteria:

* Being over 50 years or under 18 years
* Malignancy and other systemic diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with 50% Reduction of Headache Frequency | 6 months
  Monthly headache frequency will be followed

SECONDARY OUTCOMES:
Side effects | 6 months
  Major and minor side effects will be followed

CONTACTS AND LOCATIONS:
Locations (1):
- Cem Bölük, Istanbul, Fatih, Turkey (Türkiye)